CLINICAL TRIAL: NCT04444050
Title: Randomized, Double-Blind, Placebo-Controlled Single- and Multiple-Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of BMS-986331 in Healthy Participants
Brief Title: Study to Evaluate the Safety, Tolerability, Drug Levels and Drug Effects of BMS-986331 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Basic Science
Other Study IDs: CV023-005
Record Dates: First submitted 2020-06-19; First posted 2020-06-23 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Healthy Participants
Keywords: Healthy participants

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (16):
- Part 1 Single Ascending Dose (SAD): Panel 1 (Experimental)
  Interventions: Drug: BMS-986331; Other: Placebo, Matching BMS-986331
- Part 1 SAD: Panel 2 (Experimental)
  Interventions: Drug: BMS-986331; Other: Placebo, Matching BMS-986331
- Part 1 SAD: Panel 3 (Experimental)
  Interventions: Drug: BMS-986331; Other: Placebo, Matching BMS-986331
- Part 1 SAD: Panel 4 (Experimental)
  Interventions: Drug: BMS-986331; Other: Placebo, Matching BMS-986331
- Part 1 SAD: Panel 5 (Experimental)
  Interventions: Drug: BMS-986331; Other: Placebo, Matching BMS-986331
- Part 1 SAD: Panel 6 (Experimental)
  Interventions: Drug: BMS-986331; Other: Placebo, Matching BMS-986331
- Part 1 SAD: Optional Split-dose Panel (Experimental)
  Interventions: Drug: BMS-986331; Other: Placebo, Matching BMS-986331
- Part 2 Multiple Ascending Dose (MAD): Panel 1 (Experimental)
  Interventions: Drug: BMS-986331; Other: Placebo, Matching BMS-986331
- Part 2 MAD: Panel 2 (Experimental)
  Interventions: Drug: BMS-986331; Other: Placebo, Matching BMS-986331
- Part 2 MAD: Panel 3 (Experimental)
  Interventions: Drug: BMS-986331; Other: Placebo, Matching BMS-986331
- Part 2 MAD: Panel 4 (Experimental)
  Interventions: Drug: BMS-986331; Other: Placebo, Matching BMS-986331
- Part 2 MAD: Optional (to be determined) Panel (Experimental)
  Interventions: Drug: BMS-986331; Other: Placebo, Matching BMS-986331
- Part 3 MAD in Japanese Participants (J-MAD): Panel 1 (Experimental)
  Interventions: Drug: BMS-986331; Other: Placebo, Matching BMS-986331
- Part 3 J-MAD: Panel 2 (Experimental)
  Interventions: Drug: BMS-986331; Other: Placebo, Matching BMS-986331
- Part 3 J-MAD: Panel 3 (Experimental)
  Interventions: Drug: BMS-986331; Other: Placebo, Matching BMS-986331
- Part 3 J-MAD: Optional (to be determined) Panel (Experimental)
  Interventions: Drug: BMS-986331; Other: Placebo, Matching BMS-986331

INTERVENTIONS:
Drug: BMS-986331 — Specified dose on specified days
Other: Placebo, Matching BMS-986331 — Specified dose on specified days

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, drug levels and drug effects of single and multiple oral doses of BMS-986331 versus placebo in healthy participants and healthy Japanese participants.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant deviations in medical history, physical examination, ECGs, vital signs, and clinical laboratory determinations
* A body mass index of 18 - 32 kg/m2, inclusive
* Women and men must agree to follow specific methods of contraception, if applicable

For J-MAD Part 3

* Must be Japanese (both biological parents are ethnically Japanese)

Exclusion Criteria:

* Women who are of childbearing potential
* Women who are pregnant or breastfeeding
* Any significant acute or chronic medical illness
* Current or recent (within 3 months of study drug administration) gastrointestinal disease that could impact upon the absorption of study drug
* Any surgery within 12 weeks of study drug administration

Other protocol-defined inclusion/exclusion criteria apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2020-06-23 (Actual); Primary Completion 2021-05-19 (Actual); Study Completion 2021-05-19 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | Up to 13 months
Number of participants with clinical laboratory abnormalities | Up to 46 days
Number of participants with vital sign abnormalities | Up to 46 days
Number of participants with electrocardiogram (ECG) abnormalities | Up to 46 days

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) | Up to 17 days
Time to reach Cmax in plasma (Tmax) | Up to 17 days
Area under the plasma concentration-time curve from time 0 (dosing) to the time of the last quantifiable concentration observed [AUC(0-T)] | Up to 17 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- United States (2):
  - Local Institution - 0001, Anaheim, California
  - ICON (LPRA) - Lenexa, Lenexa, Kansas

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm